CLINICAL TRIAL: NCT03788889
Title: A Randomized, Double-Blinded, Placebo-Controlled Study Evaluating Phenobarbital and Ketamine Adjunctive Therapies in the Treatment of Alcohol Withdrawal Syndrome
Brief Title: Alcohol Withdrawal Syndrome Treated With Adjunctive Phenobarbital or Ketamine
Acronym: PKAT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: internal practice and policy limitations including time commitment / workflow issues
Sponsor: Santa Barbara Cottage Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-94
Record Dates: First submitted 2018-12-22; First posted 2018-12-28 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Alcohol Withdrawal Syndrome
Keywords: Lorazepam; Ketamine; Phenobarbital
MeSH Terms: interventions — Ketamine; Phenobarbital; Lorazepam; Saline Solution

STUDY DESIGN:
Intervention Model Description: prospective, randomized control trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Each participant will be randomized according to a web-based randomization program employed by a research pharmacist once the Emergency Department provider deems the patient appropriate for inpatient treatment of alcohol withdrawal syndrome.
  Each medication will be packaged by Santa Barbara Cottage Hospital pharmacy. In order to blind both the clinicians and the participants, the pharmacy will provide medication bags that are identical. Therefore, Emergency Department nursing staff and physicians will be unaware of which study drug is being provided to the patient. Normal saline will be used as a placebo to mimic study drugs (phenobarbital and ketamine). Pharmacy will remain unblinded and maintain records of which treatment assignment is prepared for each patient.
  Treatment will be provided for the duration of the patient's hospitalization; therefore, treatment compliance will be documented in the electronic health record using the medication bag identifier.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lorazepam + Ketamine + Placebo A (Active Comparator): Ketamine - infusion (0.15 - 0.4 mg/kg/hr) and placebo injections titrated by increases of 0.075 mg/kg/hr every 30 minutes for Clinical Institute Withdrawal Assessment for Alcohol (revised version) (CIWA-Ar) greater than or equal to 10 in addition to lorazepam symptom-triggered therapy
  Ketamine dosing will be based on ideal body weight
  Ketamine infusion will be discontinued once CIWA-Ar less than 10 for 4 hours
  Interventions: Drug: Ketamine; Drug: Lorazepam; Drug: Placebo A
- Lorazepam + Phenobarbital + Placebo B (Active Comparator): Phenobarbital - IV push (260 mg loading followed by 130 mg q1 hour) with placebo infusion until CIWA-Ar less than 10 with a maximum daily dose of 10mg/kg in addition to lorazepam symptom-triggered dosing for recurrent symptoms (Gold 2007)
  Maximum daily dose will be used in order to prevent over sedation as well as provide adequate storage in pharmacy monitored refrigerators for study drugs
  Interventions: Drug: Phenobarbital; Drug: Lorazepam; Drug: Placebo B
- Lorazepam + Placebo A + Placebo B (Placebo Comparator): Lorazepam will be administered every 30 minutes as indicated based on CIWA-Ar protocol for Cottage Health in addition to placebo injections and placebo infusion
  Interventions: Drug: Lorazepam; Drug: Placebo A; Drug: Placebo B

INTERVENTIONS:
Drug: Ketamine — Ketamine infusion
  Other Names: Ketalar
  Arms: Lorazepam + Ketamine + Placebo A
Drug: Phenobarbital — Phenobarbital intravenous injection
  Other Names: Solfoton, Luminal
  Arms: Lorazepam + Phenobarbital + Placebo B
Drug: Lorazepam — Standard of Care
  Other Names: Ativan
Drug: Placebo A — Placebo injection
  Other Names: Normal saline
  Arms: Lorazepam + Ketamine + Placebo A; Lorazepam + Placebo A + Placebo B
Drug: Placebo B — Placebo infusion
  Other Names: Normal saline
  Arms: Lorazepam + Phenobarbital + Placebo B; Lorazepam + Placebo A + Placebo B

SUMMARY:
The goal of this study will aim to determine if adding phenobarbital or ketamine to a symptom-triggered benzodiazepine regimen decreases the rate of intensive care unit admissions during the treatment of alcohol withdrawal syndrome when compared to symptom-triggered benzodiazepine therapy alone.

DETAILED DESCRIPTION:
The primary objective of this study is to compare phenobarbital and ketamine adjunctive therapies to lorazepam-based therapy in the treatment of acute alcohol withdrawal syndrome.

It is hypothesized that the use of an alternative agent, either phenobarbital or ketamine, when used as an adjunct to symptom-triggered lorazepam therapy will significantly reduce the rate of intensive care unit admissions and thereby reduce the total cost associated with hospital admission for treatment of alcohol withdrawal syndrome.

Enrolled patients will be admitted to Santa Barbara Cottage Hospital where they will be monitored with continuous pulse oximetry and cardiac telemetry. They will remain hospitalized while undergoing study-guided therapy in addition to supportive care for acute alcohol withdrawal syndrome. Patients will undergo standard of care therapy with lorazepam symptom-triggered therapy regardless of study participation.

ELIGIBILITY:
Inclusion Criteria:

* Primary admitting diagnosis of acute alcohol withdrawal syndrome based on International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10), code F10.3, F10.4.

Exclusion Criteria:

* Significant comorbid medical illness requiring Intensive Care Unit admission;
* Pregnancy;
* Inability to obtain intravenous access;
* Child Pugh Class C; and
* Allergy to study medications (phenobarbital, ketamine, lorazepam).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-12 (Estimated); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Intensive Care Unit admission rate | Presentation to Emergency Department through hospital stay, data will be utilized through study completion, anticipated 2 years
  Number of admissions to the intensive care unit

SECONDARY OUTCOMES:
Incidence of withdrawal seizures | Presentation to Emergency Department through hospital stay, data will be utilized through study completion, anticipated 2 years
  Number of patients with documented seizures while treated for alcohol withdrawal syndrome
Clinical Institute Withdrawal Assessment of Alcohol Scale, Revised (CIWA-Ar) scores | Presentation to Emergency Department through hospital stay, data will be utilized through study completion, anticipated 2 years
  CIWA-Ar scores (initial, maximum, discharge); Total score is cumulative of subscale measures: Minimum score is 0 (no evidence of alcohol withdrawal), Maximum score is 67 (severe alcohol withdrawal)
  Subscale measures:
  A) Nausea and vomiting (score 0-7); B) Tremor (score 0-7); C) Paroxysmal sweats (score 0-7); D) Anxiety (score 0-7); E) Tactile disturbances (score 0-7); F) Auditory disturbances (score 0-7); G) Visual disturbances (score 0-7); H) Headache, fullness in head (score 0-7); I) Agitation (score 0-7); J) Orientation and clouding of sensorium (score 0-4)
Cumulative dose of medication/s administered | Presentation to Emergency Department through hospital stay, data will be utilized through study completion, anticipated 2 years
  Cumulative dose of Lorazepam, Ketamine, and Phenobarbital
Incidence of refractory alcohol withdrawal requiring alternative sedation with dexmedetomidine, propofol or midazolam infusions | Presentation to Emergency Department through hospital stay, data will be utilized through study completion, anticipated 2 years
  Number of patients who require Dexmedetomidine, Propofol or Benzodiazepine continuous infusions and average dose while being treated for alcohol withdrawal syndrome
Rate of mechanical ventilation | Presentation to Emergency Department through hospital stay, data will be utilized through study completion, anticipated 2 years
  Rate of intubation
Incidence of alcohol withdrawal hallucinations | Presentation to Emergency Department through hospital stay, data will be utilized through study completion, anticipated 2 years
  Number of patients with documented auditory or visual hallucinations

CONTACTS AND LOCATIONS:
Overall Officials: Noah Stites-Hallet, MD, Principal Investigator — Santa Barbara Cottage Hospital

IPD SHARING:
Plan to Share IPD: No